CLINICAL TRIAL: NCT02703051
Title: A Phase 1, Open-Label Study to Evaluate the Pharmacodynamics, Safety and Tolerability of GMI-1271 With and Without Filgrastim in Healthy Adult Subjects
Brief Title: A Study to Evaluate the PK, Safety and Tolerability of GMI-1271 With and Without Filgrastim in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlycoMimetics Incorporated (Industry)
Collaborators: Celerion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: GMI-1271-103
Record Dates: First submitted 2016-03-03; First posted 2016-03-09 (Estimated); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — uproleselan; Filgrastim

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- GMI-1271 (Experimental): GMI-1271
  Interventions: Drug: GMI-1271; Drug: Placebo Injection
- Filgrastim (Active Comparator): Filgrastim
  Interventions: Drug: Filgrastim; Drug: Placebo Infusion
- GMI-1271 with Filgrastim (Experimental): GMI-1271 with Filgrastim
  Interventions: Drug: GMI-1271; Drug: Filgrastim

INTERVENTIONS:
Drug: GMI-1271
  Arms: GMI-1271; GMI-1271 with Filgrastim
Drug: Filgrastim
  Arms: Filgrastim; GMI-1271 with Filgrastim
Drug: Placebo Injection
  Arms: GMI-1271
Drug: Placebo Infusion
  Arms: Filgrastim

SUMMARY:
Phase 1, open-label, parallel, active-controlled, multiple IV dose, proof of concept study conducted at one study center in the United States (US).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male and/or females, 19 to 60 years of age, inclusive.
2. Medically healthy with no clinically significant screening results as deemed by the PI.

Exclusion Criteria:

1. History of presence of clinically significant medical condition or disease in the opinion of the PI.
2. Alcoholism or drug abuse.
3. Liver disease.
4. Female subjects who are pregnant or lactating.
5. Known history or evidence of active hepatitis A, B, or C or HIV.
6. Clinically significant cardiovascular disease.
7. Participation in another clinical trial within 28 days prior to the first dose of GMI-1271 or filgrastim, whichever occurs first.

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Measurement of subsets of WBC | 10 days

SECONDARY OUTCOMES:
Number of adverse events as a measure of safety and tolerability | 19 days

CONTACTS AND LOCATIONS:
Overall Officials: Laura Sterling, MD, Principal Investigator — Celerion
Locations (1):
- Celerion, Lincoln, Nebraska, United States